CLINICAL TRIAL: NCT02973269
Title: A Phase 2, Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial of DaxibotulinumtoxinA for Injection for the Management of Plantar Fasciitis
Brief Title: DaxibotulinumtoxinA for Injection for the Management of Plantar Fasciitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New trial with same indication initiated
Sponsor: Revance Therapeutics, Inc. (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT002-CL008
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAXI 240 U (Experimental): DaxibotulinumtoxinA for injection for the treatment of plantar fasciitis (PF) with 240 U
  Interventions: Biological: daxibotulinumtoxin type A
- Placebo (Placebo Comparator): Placebo Intramuscular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: daxibotulinumtoxin type A — Intramuscular injection
  Other Names: DAXI
  Arms: DAXI 240 U
Biological: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
The specific aim of the study is to compare the safety and efficacy of a single administration of DaxibotulinumtoxinA for Injection versus placebo for managing plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, including authorization to release health information
* Skeletally mature, male or female patients 18 to 65 years of age with diagnosis of plantar fasciitis
* Persistent heel pain for more than three months
* Women of child bearing potential must have a negative urine pregnancy test (UPT) at Screening Visit and must use an effective method of birth control during the course of the study

Exclusion Criteria:

* Previous surgery on the midfoot or hindfoot
* Neuromuscular disease
* Systemic muscle weakness
* Planning a pregnancy during the study
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to first visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo group
Period: Overall Study
Arm/Group | DAXI 240 U | Placebo
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | DAXI 240 U | Placebo | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
AOFAS total score [Mean (Standard Deviation); unit: units on a scale] | 71.3 (2.5) | 66.0 (21.7) | 68.3 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the American Orthopaedic Foot and Ankle Score (AOFAS)
Description: The American Orthopaedic Foot and Ankle Score (AOFAS) is a 9-item questionnaire that evaluates pain, function, and alignment of the foot and ankle. The total score ranges from 0 to 100, with lower scores representing greater pain and disability, and higher scores representing better function.
Time Frame: 16 weeks
Population: The Intent-to-Treat population includes all patients randomized to treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DAXI 240 U | Placebo
Number analyzed (Participants) | 3 | 4
units on a scale | 81.3 (11.0) | 86.5 (12.1)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs
Arm/Group | DAXI 240 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 240 U (N=3) | Placebo (N=4)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (45) days prior to the submission thereof for publication or disclosure to a third party:(i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT02973269/Prot_SAP_000.pdf